CLINICAL TRIAL: NCT04207580
Title: A National Prospective Cohort of Patients With Idiopathic Nephrotic Syndrome Beginning in Childhood.
Acronym: PIN'SNP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0006
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Idiopathic Nephrotic Syndrome
Keywords: Cohort - Idiopathic nephrotic syndrome - child
MeSH Terms: conditions — Nephrosis, Lipoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, hair and nails will be collected at the beginning of the NIS (before starting immunosuppressive treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inclusion and follow up of pediatric patients: Inclusion and follow up of pediatric patients with an idiopathic nephrotic syndrome, from the beginning of the disease to 18 years old or transfer of the follow-up to a nephrology unit for adults.
  130 new patients are expected to be included on an annual basis.
  Interventions: Other: Inclusion and follow up of pediatric patients with an idiopathic nephrotic syndrome,

INTERVENTIONS:
Other: Inclusion and follow up of pediatric patients with an idiopathic nephrotic syndrome, — The study consists in collecting clinical, biological, psychological and social data of INS pediatric patients.
  A bio collection is also created: blood, urine, hair and nails will be collected at the beginning of the INS (before starting immunosuppressive treatment).

SUMMARY:
Pediatric idiopathic nephrotic syndrome (INS) is a rare disease for which the optimal therapeutic strategy has not yet been defined. A network of clinicians treating complicated forms of this disease (grouped within the Société de Néphrologie Pédiatrique, SNP) exists, but to date there is no prospective cohort following up these patients that would facilitate the development of cohort-nested trials. This absence of structured follow up makes it difficult to set up prospective studies.

The main objective is to create a prospective cohort of pediatric INS patients to collect cases treated in SNP centers, to study their epidemiological characteristics, and to provide a basis for comparison for future cohort-nested trials.

DETAILED DESCRIPTION:
In this study, data from patients with INS will be recorded prospectively, regularly and systematically. The cohort will be composed of patients followed by pediatric nephrologists affiliated with the SNP. Metropolitan France, Reunion Island and Mayotte are the geographical areas concerned. It is planned to integrate other French overseas departments and territories, in particular the West Indies.

This is therefore a prospective, multicenter, cohort follow-up study. The data will be centralized via a secure website dedicated to the study.

Data will be obtained from:

* Medical record data (hospitalization/consultations) as part of routine clinical follow-up for patients with active disease. This information will be medically validated and integrated into the database with the help of clinical research staff.
* A telephone interview for annual follow-ups for patients whose absence of active disease no longer requires a systematic medical visit. This structured interview will be administered by telephone by the study's clinical research staff.
* Self-administered or hetero-administered quality of life questionnaires (PEDS-QL), self-administered or hetero-administered treatment compliance questionnaires (Morisky's Score), and questionnaires on the aesthetic impact of treatments (Ferriman's Score). These questionnaires will be centralized and reported to the database by the study's clinical research staff.

ELIGIBILITY:
Inclusion Criteria:

* Patient under 18 years of age
* With idiopathic nephrotic syndrome (according to SPN criteria) beginning after January 1, 2018
* Child seen at least once in consultation or hospitalization by a pediatrician member of the Society of Pediatric Nephrology
* Residing in France
* Consent signed by parents and patient's agreement to participate (if of age)
* Affiliated to a social security system.

Exclusion Criteria:

* Refusal of the patient or legal representatives to participate in the cohort

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric idiopathic nephrotic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2045-01 (Estimated)

PRIMARY OUTCOMES:
Number of cases included in the cohort and description of their characteristics | 2 years
  * Number of followed cases, gender, and age
  * Geographical localization of followed cases
  * Progressive disease pattern (relapses, corticosteroid dependence, other treatments used)
  * Serious side effects related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Guigonis, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Limoges Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahans C, Boyer O, Dunand O, Parmentier C, Ranchin B, Roussey G, Samaille C, Tellier S, Vrillon I, Preka E, Meriguet T, Dubrasquet A, Ichay L, Clave S, Bernardor J, Merieau E, Dossier C, Guigonis V. A "Trial within a Cohort" platform for pediatric clinical trials on idiopathic nephrotic syndrome: scope, objectives, and design of the retrospective-prospective cohort PIN'SNP. Pediatr Nephrol. 2025 Jul;40(7):2225-2238. doi: 10.1007/s00467-025-06676-7. Epub 2025 Mar 3. PMID 40032676